CLINICAL TRIAL: NCT04951245
Title: Ultrasound-assisted Carbon Nanoparticle Suspensions Mapping Versus Dual-tracer-guided Sentinel Lymph Node Biopsy in Patients With Early Breast Cancer (UltraCars): a Prospective, Randomized Controlled Phase 3 Trial
Brief Title: Ultrasound-assisted CNSs Mapping Versus Dual-tracer-guided Sentinel Lymph Node Biopsy
Acronym: UltraCars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190511
Record Dates: First submitted 2019-09-21; First posted 2021-07-06 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UC group (Experimental): Ultrasound-assisted CNSs guided SLN mapping
  Interventions: Procedure: UC group: ultrasound-assisted CNSs guided
- GC group (Active Comparator): CNSs plus ICG dual-tracer-guided SLN mapping
  Interventions: Procedure: GC group: CNSs plus ICG dual-tracer-guided

INTERVENTIONS:
Procedure: UC group: ultrasound-assisted CNSs guided — 1ml of CNSs was subcutaneously injected into the areolar area in the upper outer quadrant of the breast. The injection site was massaged for 15 minutes to promote drainage of the tracer to the axilla. During the intraoperative ultrasound-assisted procedure, an ultrasound diagnostic system was used. Before the incision, ultrasound-guided exploration of SLNs was performed by placing the probe on the lateral border of the breast and sliding cranially along the lateral border of the pectoralis major muscle . A sterile skin marker was then used to mark the optimal site of incision over the targeted lymph nodes, and the distance from the skin to the nodes was measured by ultrasound and recorded in millimeters. Blunt dissection was carried out to identify the CNSs-stained nodes around the marked region. Ultrasonography probe was placed repeatedly in or around the wound at different angles for adequate visualization if SLNs could not be localized with further dissection.
  Arms: UC group
Procedure: GC group: CNSs plus ICG dual-tracer-guided — The preparation of CNSs mapping was identical to that of the UC group. 1ml of diluted ICG was subsequently injected into the areolar area in the upper outer quadrant of the breast. A NIR camera was used to visualize the subcutaneous lymph vessels and localized the SLNs. All fluorescent or black-stained lymph nodes along with any palpable suspicious nodes were removed. The remaining surgical field was reexamined to ensure complete resection of fluorescent lymph nodes.
  Arms: GC group

SUMMARY:
The investigators suggested ultrasound-assisted Carbon nanoparticle suspensions (CNSs) mapping had great clinical value in clinical application and might serve as a useful alternative to the dual-tracer-guided SLNB. The investigators designed this prospective, randomized controlled phase 3 trial, to compare the feasibility and diagnostic performance of ultrasound-assisted carbon nanoparticle suspensions mapping versus dual-tracer-guided sentinel lymph node biopsy in patients with early breast cancer.

DETAILED DESCRIPTION:
The study was a single-center, open-label, randomized controlled, non-inferiority, phase 3 trial. Eligible participants were 18 year's of age or older and had histologically confirmed primary invasive breast cancer, or ductal carcinoma in situ scheduled for mastectomy, without clinical or radiological nodal involvement (cN0) or with clinical positive lymph nodes (cN1) that were downstaged to cN0 following neoadjuvant chemotherapy (NCT); and had an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1. Participants were randomly assigned (1:1) using a permuted block randomization scheme to receive either ultrasound-assisted CNSs (UC group) or CNSs plus ICG dual-tracer-guided (GC group) SLN mapping.

ELIGIBILITY:
Inclusion criteria:

1. The participants must be female and 18 years of age or older.
2. Resectable invasive adenocarcinoma of the breast, confirmed histologically.
3. Ductal carcinoma in situ confirmed histologically.
4. The participants must be a preoperative clinical Tis, T1, T2, T3 as well as clinical M0 breast cancer.
5. Without clinical or radiological nodal involvement (cN0): No positive ipsilateral axillary lymph nodes; No prior removal of ipsilateral axillary lymph nodes; No suspicious palpable nodes in the contralateral axilla or palpable supraclavicular or infraclavicular nodes, unless proven nonmalignant by biopsy.
6. With clinical positive lymph nodes (cN1) (including any abnormal or enlarged clinically palpable lymph nodes or core biopsy/surgical biopsy/FNA evidence of malignant cell within any lymph nodes) that was downstaged to cN0 following neoadjuvant therapy.
7. The participants must have an ECOG performance status of Grade 0-1.
8. The participants must provide written informed consent before participating in the study.

Exclusion criteria:

1. The breast has ulceration, erythema, infiltration of the skin or underlying chest wall (complete fixation), peau d'orange, or skin edema of any magnitude. Tethering or dimpling of the skin or nipple inversion allowed.
2. The participants has a known hypersensitivity to tracers planned for use during SLNB.
3. Other prior breast malignancy except lobular carcinoma in situ.
4. The participants has had prior breast implants.
5. The participants has had prior breast reduction surgery.
6. The participants has had other prior surgery in the upper, outer quadrant, areola, or axilla to the indicated breast.
7. The participants has a positive pregnancy test or is lactating.
8. The participants has participated in another investigational drug study during the 30 days prior to signing informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
The identification rate of SLNs | within 14 days of SLNB
  Defined as the number of patients who at least one SLN were detected divided by the total number of patients included.

SECONDARY OUTCOMES:
The mean number of SLNs collected | within 14 days of SLNB
  Defined as the number of tracer-stained or palpable SLNs divided by the number of patients whose SLNs were identified.
Operative time | within 14 days of SLNB
  Defined as the time from skin incision to resection of the SLNs specimens in patients whose at least one SLN were detected.
Intraoperative or postoperative complications | within 30 days of SLNB
  An adverse event is any untoward, undesired, and/or unplanned clinical event in the form of signs, symptoms, disease, or laboratory testing, or physiological observations occurring in a human participating in a clinical study with a study drug, regardless of causal relationship.

OTHER OUTCOMES:
Identification rate of SLNs in post-NCT patients | within 14 days of SLNB
  Defined as the number of patients who at least one SLN were detected divided by the total number of patients included in NCT subgroup.

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, China

REFERENCES:
- [Derived] Zhang L, Cheng M, Lin Y, Zhang J, Shen B, Chen Y, Yang C, Yang M, Zhu T, Gao H, Ji F, Li J, Wang K. Ultrasound-assisted carbon nanoparticle suspension mapping versus dual tracer-guided sentinel lymph node biopsy in patients with early breast cancer (ultraCars): phase III randomized clinical trial. Br J Surg. 2022 Nov 22;109(12):1232-1238. doi: 10.1093/bjs/znac311. PMID 36074703